CLINICAL TRIAL: NCT04210115
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Trial of Pembrolizumab (MK-3475) Versus Placebo in Participants With Esophageal Carcinoma Receiving Concurrent Definitive Chemoradiotherapy (KEYNOTE 975)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Placebo in Participants With Esophageal Carcinoma Who Are Receiving Chemotherapy and Radiation Therapy (MK-3475-975/KEYNOTE-975)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-975; MK-3475-975 (Other: MSD); KEYNOTE-975 (Other: MSD); PHRR200210-002490 (Registry Identifier: PHRR); 205261 (Registry Identifier: Japic-CTI); 2022-501531-16 (Registry Identifier: EU CT); 2019-002006-51 (EudraCT Number)
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); Gastroesophageal Junction Carcinoma (GEJC); Esophageal Adenocarcinoma (EAC)
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Death-Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Saline Solution; Cisplatin; Fluorouracil; Radiotherapy; Leucovorin; Levoleucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+FP or FOLFOX Therapy+Radiotherapy (Experimental): Participants receive pembrolizumab 200 mg on Day 1 of each 3-week cycle for 8 cycles followed by pembrolizumab 400 mg on Day 1 of each 6-week cycle for 5 cycles PLUS either:
  * FP therapy: cisplatin 75 mg/m^2 on Day 1 of Weeks 1, 5, 8 and 11 PLUS 5-fluorouracil (5-FU)] 1000 mg/m^2 per day on Days 1-4 of Weeks 1, 5, 8 and 11 OR 800 mg/m^2/day on each of Days 1-5 at Weeks 1, 5, 8, and 11 PLUS radiotherapy (either 50 Gray [Gy] in 25 fractions OR 60 Gy in 30 fractions) on Days 1-5 of each 3-week cycle OR
  * FOLFOX therapy: oxaliplatin 85 mg/m^2 AND either leucovorin 400 mg/m^2 OR levoleucovorin 200 mg/m^2 on Day 1 of Weeks 1, 3, 5, 7, 9 and 11 PLUS either 5-FU 400 mg/m^2 on Day 1 of Weeks 1, 3, 5, 7, 9 and 11 OR 5-FU 800 mg/m^2 per day on Days 1 and 2 of Weeks 1, 3, 5, 7, 9 and 11 PLUS radiotherapy (50 Gy in 25 fractions) on Days 1-5 of each 3-week cycle.
  All treatments except radiotherapy are given by intravenous (IV) infusion. Total treatment duration is approximately 1 year.
  Interventions: Biological: pembrolizumab; Drug: cisplatin; Drug: 5-FU; Radiation: radiotherapy; Drug: leucovorin; Drug: levoleucovorin; Drug: oxaliplatin
- Placebo+FP or FOLFOX Therapy+Radiotherapy (Placebo Comparator): Participants receive placebo on Day 1 of each 3-week cycle for 8 cycles followed by placebo on Day 1 of each 6-week cycle for 5 cycles PLUS either:
  * FP therapy: cisplatin 75 mg/m^2 on Day 1 of Weeks 1, 5, 8 and 11 PLUS 5-FU 1000 mg/m^2 per day on Days 1-4 of Weeks 1, 5, 8 and 11 OR 800 mg/m^2/day on each of Days 1-5 at Weeks 1, 5, 8, and 11 PLUS radiotherapy (either 50 Gy in 25 fractions OR 60 Gy in 30 fractions) on Days 1-5 of each 3-week cycle OR
  * FOLFOX therapy: oxaliplatin 85 mg/m^2 AND either leucovorin 400 mg/m^2 OR levoleucovorin 200 mg/m^2 on Day 1 of Weeks 1, 3, 5, 7, 9 and 11 PLUS either 5-FU 400 mg/m^2 on Day 1 of Weeks 1, 3, 5, 7, 9 and 11 OR 5-FU 800 mg/m^2 per day on Days 1 and 2 of Weeks 1, 3, 5, 7, 9 and 11 PLUS radiotherapy (50 Gy in 25 fractions) on Days 1-5 of each 3-week cycle.
  All treatments except radiotherapy are given by IV infusion. Total treatment duration is approximately 1 year.
  Interventions: Drug: placebo; Drug: cisplatin; Drug: 5-FU; Radiation: radiotherapy; Drug: leucovorin; Drug: levoleucovorin; Drug: oxaliplatin

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+FP or FOLFOX Therapy+Radiotherapy
Drug: placebo — IV infusion
  Other Names: Normal saline solution
  Arms: Placebo+FP or FOLFOX Therapy+Radiotherapy
Drug: cisplatin — IV infusion
  Other Names: PLATINOL®
Drug: 5-FU — IV infusion
  Other Names: ADRUCIL®
Radiation: radiotherapy — external radiation
Drug: leucovorin — IV infusion
  Other Names: calcium folinate; folinic acid
Drug: levoleucovorin — IV infusion
  Other Names: FUSILEV®; calcium levofolinate; levofolinic acid
Drug: oxaliplatin — IV infusion
  Other Names: ELOXATIN®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of treatment with definitive chemoradiotherapy (dCRT) + pembrolizumab (MK-3475) compared to treatment with dCRT + placebo with respect to Event-free Survival (EFS) and Overall Survival (OS) in:

* participants whose tumors express Programmed Death-Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10
* participants whose tumors express PD-L1 CPS ≥1
* all participants

The primary study hypotheses are that dCRT+ pembrolizumab is better than dCRT + placebo with respect to:

* EFS in participants whose tumors express PD-L1 CPS ≥10
* EFS in participants whose tumors express PD-L1 CPS ≥1
* EFS in all participants
* OS in participants whose tumors express PD-L1 CPS ≥10
* OS in participants whose tumors express PD-L1 CPS ≥1
* OS in all participants

DETAILED DESCRIPTION:
Participants receive pembrolizumab or placebo PLUS one of two chemotherapy regimens PLUS radiation therapy for up to approximately one year. The chemotherapy regimens are either:

* FP (5-fluorouracil [5-FU] + cisplatin) or
* FOLFOX (5-FU + oxaliplatin + leucovorin or levoleucovorin).

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of CTX N+ M0 or cT2-T4a NX M0 ESCC, GEJC, EAC, or histologically or cytologically confirmed diagnosis of cTX N+ M1 cervical or upper thoracic esophageal carcinoma with supraclavicular lymph node metastases only
* Is deemed suitable for dCRT
* Is ineligible for curative surgery based on the documented opinion of a qualified medical/surgical/radiation oncologist.
* Is not expected to require tumor resection during the course of the study
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 3 days of the first dose of study treatment
* Has adequate organ function
* Male participants must use adequate contraception (a male condom plus partner use of an additional contraceptive method) unless confirmed to be azoospermic (vasectomized or secondary to medical cause) and refrain from donating sperm during the study treatment period and through 90 days after the last dose of chemotherapy
* Female participants who are a Woman of Childbearing Potential (WOCBP) must use contraception that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle, during the study treatment period through 180 days after the last dose of chemotherapy or 120 days after the last dose of pembrolizumab, whichever is greater, and agree not to donate eggs to others or freeze/store for her own use for the purpose of reproduction during this period
* Female participants must not be pregnant or breastfeeding

Exclusion Criteria:

* Has direct invasion of tumor into adjacent organs such as the aorta or trachea or has radiographic evidence of >90 degree encasement or invasion of a major blood vessel, or of intratumoral cavitation
* Has had major surgery other than for insertion of a feeding tube, open biopsy, or significant traumatic injury within 28 days prior to randomization, or anticipates the need for major surgery during study treatment; participants with gastric or esophageal fistulae are excluded
* Has had weight loss of >20% in the previous 3 months
* Has had prior chemotherapy or radiotherapy for esophageal cancer
* Has had a myocardial infarction within the past 6 months
* Has symptomatic congestive heart failure
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-programmed cell death-ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention; administration of killed vaccines is allowed
* Has received any prior systemic anticancer therapy for esophageal cancer including investigational agents
* Has not recovered from all adverse events (AEs) due to previous non-anticancer therapies to ≤Grade 1 or Baseline
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded from the study. Participants with localized prostate cancer that has undergone potentially curative treatment can be enrolled in the study.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, any of the study chemotherapy agents, or their excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment (180 days for participants receiving cisplatin who are breastfeeding)
* Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) | Up to ~60 months
  EFS is defined as the time from randomization to an event defined as local, regional, or distant radiological recurrence as assessed by the investigator; clinical recurrence as assessed by the investigator with histopathologic confirmation (in the absence of radiological disease recurrence by investigator assessment); or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to ~72 months
  OS is defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Number of participants with an adverse event (AE) | Up to ~15 months
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants discontinuing study treatment due to an adverse event (AE) | Up to ~12 months
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (170):
- United States (19):
  - MemorialCare Health System - Long Beach Medical Center-Oncology ( Site 0691), Long Beach, California
  - Columbus Regional Research Institute ( Site 0047), Columbus, Georgia
  - University of Kansas Cancer Center ( Site 0023), Westwood, Kansas
  - Cancer Center of Kansas ( Site 0058), Wichita, Kansas
  - University Medical Center ( Site 0035), New Orleans, Louisiana
  - Greater Baltimore Medical Center ( Site 0031), Baltimore, Maryland
  - Dana Farber Cancer Center ( Site 0034), Boston, Massachusetts
  - Henry Ford Hospital ( Site 0685), Detroit, Michigan
  - University of Missouri ( Site 0688), Columbia, Missouri
  - Renown Regional Medical Center ( Site 0706), Reno, Nevada
  - Rutgers Cancer Institute of New Jersey ( Site 0695), New Brunswick, New Jersey
  - Weill Cornell Medical College ( Site 0053), New York, New York
  - Stephenson Cancer Center ( Site 0044), Oklahoma City, Oklahoma
  - Oregon Health & Science University Center for Health & Healing 2- CHH2 ( Site 0060), Portland, Oregon
  - Allegheny Health Network ( Site 0042), Pittsburgh, Pennsylvania
  - Thompson Cancer Survival Center ( Site 0696), Knoxville, Tennessee
  - Utah Cancer Specialists ( Site 0697), Salt Lake City, Utah
  - Cancer Care Northwest - Spokane Valley ( Site 0036), Spokane Valley, Washington
  - University of Wisconsin Hospital and Clinics ( Site 0033), Madison, Wisconsin
- Argentina (4):
  - Instituto Medico Alexander Fleming ( Site 0063), Buenos Aires, Buenos Aires F.D.
  - Fundacion Favaloro ( Site 0061), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Hospital Municipal de Gastroenterologia Dr. Bonorino Udaondo ( Site 0066), Buenos Aires
  - CEMIC ( Site 0064), Buenos Aires
- Belgium (4):
  - UCL Saint Luc ( Site 0162), Brussels, Bruxelles-Capitale, Region de
  - UZ Gent ( Site 0163), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0161), Leuven, Vlaams-Brabant
  - AZ Delta ( Site 0165), Roeselare, West-Vlaanderen
- Brazil (4):
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 0088), Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao ( Site 0087), Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia Reichow ( Site 0085), Blumenau, Santa Catarina
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0081), São Paulo
- Canada (6):
  - Cross Cancer Institute ( Site 0010), Edmonton, Alberta
  - CancerCare Manitoba ( Site 0002), Winnipeg, Manitoba
  - The Ottawa Hospital - Cancer Care ( Site 0008), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 0012), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0011), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0005), Montreal, Quebec
- Chile (4):
  - Centro de Cancer Nuestra Senora de la Esperanza ( Site 0104), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0106), Temuco, Región de la Araucanía
  - Centro de Investigacion y desarrollo Oncologico SpA - CIDO SpA ( Site 0103), Temuco, Región de la Araucanía
  - Hospital Regional de Concepcion ( Site 0105), Concepción, Región del Biobío
- China (18):
  - Anhui Provincial Hospital-Oncology Radiotherapy Department ( Site 0531), Hefei, Anhui
  - The 900th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army ( Si, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 0538), Xiamen, Fujian
  - Hubei Cancer Hospital ( Site 0514), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0515), Changsha, Hunan
  - Huai an First People s Hospital ( Site 0526), Huai'an, Jiangsu
  - Jiangsu Cancer Hospital ( Site 0519), Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University ( Site 0522), Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University ( Site 0524), Zhenjiang, Jiangsu
  - Jiangxi Cancer Hospital ( Site 0512), Nanchang, Jiangxi
  - Shanghai Chest Hospital ( Site 0501), Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital ( Site 0503), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 0502), Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital ( Site 0527), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0505), Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital ( Site 0530), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 0523), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0529), Hangzhou, Zhejiang
- Czechia (4):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 0721), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava-Klinika onkologicka ( Site 0719), Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 0720), Olomouc, Olomoucký kraj
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 0718), Prague, Praha 5
- Denmark (2):
  - Rigshospitalet ( Site 0199), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 0200), Odense, Region Syddanmark
- Estonia (2):
  - SA Pohja-Eesti Regionaalhaigla ( Site 0201), Tallinn, Harju
  - SA Tartu Ulikooli Kliinikum ( Site 0202), Tartu, Tartu
- France (10):
  - Institut De Cancerologie De Lorraine ( Site 0222), Vandœuvre-lès-Nancy, Ain
  - Centre Francois Baclesse ( Site 0236), Caen, Calvados
  - Centre Georges Francois Leclerc ( Site 0223), Dijon, Cote-d Or
  - CHU Limoges Hopital Dupuytren ( Site 0225), Limoges, Haute-Vienne
  - Institut Curie - Centre Rene Huguenin ( Site 0237), Saint-Cloud, Hauts-de-Seine
  - Institut Jean Godinot ( Site 0238), Reims, Marne
  - CHU Hotel Dieu Nantes ( Site 0230), Nantes, Pays de la Loire Region
  - Institut Sainte Catherine ( Site 0228), Avignon, Provence-Alpes-Côte d'Azur Region
  - CHU Amiens Picardie Site Sud Amiens ( Site 0235), Amiens, Somme
  - CHD Vendee ( Site 0227), La Roche-sur-Yon, Vendee
- Germany (6):
  - Marienhospital Stuttgart Vincenz von Paul Kliniken gGmbH ( Site 0253), Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Koeln ( Site 0251), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Muenster ( Site 0248), Münster, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz ( Site 0247), Mainz, Rhineland-Palatinate
  - Charite Campus Virchow Klinikum ( Site 0250), Berlin
  - Facharztzentrum Eppendorf ( Site 0242), Hamburg
- Guatemala (6):
  - Centro de Investigaciones Clinicas de Latinoamerica S.A. - CELAN ( Site 0122), Guatemala City
  - Gastrosoluciones ( Site 0126), Guatemala City
  - Oncomedica ( Site 0125), Guatemala City
  - Grupo Medico Angeles ( Site 0121), Guatemala City
  - Medi-K Cayala ( Site 0124), Guatemala City
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 0123), Quetzaltenango
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital ( Site 0543), Hong Kong
  - Princess Margaret Hospital. ( Site 0542), Hong Kong
  - Queen Mary Hospital ( Site 0541), Pokfulam
- Hungary (4):
  - Pecsi Tudomanyegyetem AOK ( Site 0265), Pécs, Baranya
  - Bekes Megyei Kozponti Korhaz - Pandy Kalman Tagkorhaza ( Site 0262), Gyula, Bekes County
  - Orszagos Onkologiai Intezet ( Site 0263), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0261), Debrecen
- Italy (9):
  - Fondazione IRCCS Policlinico San Matteo-Oncology ( Site 0300), Pavia, Lombardy
  - IRCCS Policlinico San Donato ( Site 0295), San Donato Milanese, Milano
  - Azienda Ospedaliero Universitaria Pisana - Presidio Santa Chiara ( Site 0294), Pisa, Tuscany
  - ASST Papa Giovanni XXIII ( Site 0296), Bergamo
  - Azienda Socio Sanitaria Territoriale di Cremona ( Site 0299), Cremona
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0292), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-SC Oncologia Clinica Sperimentale Addome ( Site 0, Napoli
  - IRCCS Istituto Oncologico Veneto ( Site 0298), Padua
  - Policlinico Universitario A. Gemelli ( Site 0297), Roma
- Japan (6):
  - Aichi Cancer Center Hospital ( Site 0563), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0562), Kashiwa, Chiba
  - Kanagawa Cancer Center ( Site 0565), Yokohama, Kanagawa
  - Saitama Cancer Center ( Site 0564), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0566), Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 0561), Tokyo
- Mexico (2):
  - Cryptex Investigación Clínica S.A. de C.V. ( Site 0729), Cuauhtémoc, Ciudad de México, Mexico City
  - CENTRO HEMATO ONCOLOGICO PRIVADO-CHOP ( Site 0728), Toluca
- Peru (4):
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 0141), Lima, Muni Metro de Lima
  - Detecta Clínica ( Site 0146), Surquillo, Muni Metro de Lima
  - Hospital Nacional Arzobispo Loayza ( Site 0143), Lima
  - Clinica San Gabriel ( Site 0142), Lima
- Philippines (4):
  - Baguio General Hospital and Medical Center ( Site 0603), Baguio City, Benguet
  - Cebu Doctors University Hospital ( Site 0604), Cebu City, Cebu
  - The Medical City-Iloilo ( Site 0602), Iloilo City, Iloilo
  - St. Luke s Medical Center ( Site 0601), Quezon City, National Capital Region
- Portugal (5):
  - Hospital Beatriz Angelo ( Site 0374), Loures, Lisbon District
  - Inst. Portugues de Oncologia de Lisboa Francisco Gentil EPE ( Site 0372), Lisbon
  - Hospital da Luz ( Site 0373), Lisbon
  - CHLN Hospital Santa Maria ( Site 0376), Lisbon
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 0371), Porto
- Romania (7):
  - MedEuropa Bucuresti - Centru de Radioterapie-Oncology ( Site 0400), Bucharest, București
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 0392), Cluj-Napoca, Cluj
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 0391), Cluj-Napoca, Cluj
  - Ovidius Clinical Hospital OCH-Oncology and Hematology ( Site 0393), Ovidiu, Constanța County
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 0394), Craiova, Dolj
  - Centrul Medical Topmed ( Site 0398), Târgu Mureş, Mureș County
  - S.C.Focus Lab Plus S.R.L ( Site 0395), Bucharest
- Russia (9):
  - GBUZ Republican Clinical Oncological Dispensary-Antitumor drug therapy department ( Site 0430), Ufa, Baskortostan, Respublika
  - Kaluga Regional Clinical Oncology Center ( Site 0424), Kaluga, Kaluzskaja Oblast
  - Main Military Clinical Hospital n.a. N.N.Burdenko ( Site 0421), Moscow, Moscow
  - FSAI Treatment and Rehabilitation Centre of the MoH and SD of RF ( Site 0429), Moscow, Moscow
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 0420), Samara, Samara Oblast
  - Pavlov First Saint Petersburg State Medical University ( Site 0426), Saint Petersburg, Sankt-Peterburg
  - Medical institute named after Berezin Sergey ( Site 0417), Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Oncology Hospital ( Site 0411), Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 0412), Kazan', Tatarstan, Respublika
- South Korea (6):
  - Chonnam National University Hwasun Hospital ( Site 0625), Hwasun Gun, Jeonranamdo
  - National Cancer Center ( Site 0626), Goyang-si, Kyonggi-do
  - Asan Medical Center ( Site 0623), Songpagu, Seoul
  - Severance Hospital Yonsei University Health System ( Site 0624), Seoul
  - Samsung Medical Center ( Site 0622), Seoul
  - Korea University Guro Hospital ( Site 0621), Seoul
- Taiwan (7):
  - Chang Gung Med Foundation. Kaohsiung Branch ( Site 0643), Kaohsiung City
  - China Medical University Hospital ( Site 0646), Taichung
  - Taichung Veterans General Hospital-Radiation Oncology ( Site 0647), Taichung
  - National Cheng Kung University Hospital ( Site 0645), Tainan
  - National Taiwan University Hospital ( Site 0641), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 0644), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0642), Taoyuan District
- Turkey (Türkiye) (5):
  - Istanbul University Cerrahpasa Medical Faculty ( Site 0452), Istanbul, Istanbul
  - Memorial Ankara Hastanesi ( Site 0461), Ankara
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 0451), Istanbul
  - Ege Universitesi Tip Fakultesi ( Site 0457), Izmir
  - Izmir Katip Celebi Universitesi Ataturk Egitim ve Arastirma Hastanesi ( Site 0458), Izmir
- United Kingdom (10):
  - Aberdeen Royal Infirmary ( Site 0474), Aberdeen, Aberdeen City
  - Cambridge University Hospitals NHS Trust ( Site 0477), Cambridge, Cambridgeshire
  - Royal Free Hospital ( Site 0702), London, England
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 0283), London, London, City of
  - Hammersmith Hospital-Medical Oncology ( Site 0471), London, London, City of
  - Nottingham University Hospitals NHS Trust ( Site 0476), Nottingham, Nottinghamshire
  - Royal Marsden Hospital (Sutton) ( Site 0281), Sutton, Surrey
  - University College Hospital NHS Foundation Trust ( Site 0701), London, Worcestershire
  - The Christie NHS Foundation Trust ( Site 0282), Manchester
  - Mount Vernon Hospital ( Site 0478), Northwood

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Shah MA, Bennouna J, Doi T, Shen L, Kato K, Adenis A, Mamon HJ, Moehler M, Fu X, Cho BC, Bordia S, Bhagia P, Shih CS, Desai A, Enzinger P. KEYNOTE-975 study design: a Phase III study of definitive chemoradiotherapy plus pembrolizumab in patients with esophageal carcinoma. Future Oncol. 2021 Apr;17(10):1143-1153. doi: 10.2217/fon-2020-0969. Epub 2021 Feb 3. PMID 33533655
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26217&tenant=MT_MSD_9011